CLINICAL TRIAL: NCT04947696
Title: Towards Precision Medicine in Pancreatic Surgery - an Integrative Approach Combining Deep Learning, Genetics and Epigenetics
Brief Title: Circulating Epigenetics in Pancreatic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Martin Sillesen, MD, PhD, Assoc. Prof., Rigshospitalet, Denmark
Other Study IDs: 70711
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood cells and plasma from patients undergoing a Whipples procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients undergoing a Whipples procedure for pancreatic cancer
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Blood sampling preoperatively and sequentially up to 30 days post op

SUMMARY:
The overall objective of the study is to assess DNA-methylation changes in circulating blood cells and cell free DNA in plasma from patients undergoing the Whipples procedure for pancreatic caner

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic cancer scheduled for the Whipples procedure

Exclusion Criteria:

* Under 18 years of age
* Pregnancy
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in DNA-methylation patterns from the pre to postoperative setting | Up to 30 days postoperatively

SECONDARY OUTCOMES:
Occurence of a postoperative complication | 30 days postoperatively
Relapse of pancreatic cancer | 2 years from time of operation

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No